CLINICAL TRIAL: NCT07138365
Title: Clinical and Biochemical Effects Of Different Cryotherapy Protocols On Endodontic Treated Mandibular Premolars With Symptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Clinical and Biochemical Effects Of Cryotherapy Protocols On Mandibular Premolars With Symptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 943
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain; Inflammation
Keywords: Cryotherapy; post operative pain; inflammation; analgesic intake
MeSH Terms: conditions — Pain, Postoperative; Inflammation | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: randomized, controlled, single-blinded, single- center clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: 1)Patients will be assigned at random to either the intra oral group ,intra radicular group or the control group (n=10). The name of the group will be scrawled on a slip of paper and sealed inside a plain envelope. As each patient arrived for treatment, one envelope will be drawn at random from a box to assign the patient to a certain group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): No application of cryotherapy .Patients will receive conventional root canal treatment. Canals will be irrigated with room temperature 2.5% NaOCl. Final flush will be done with room temperature saline for 10 min.
- Oral Cryo Group (Active Comparator): custom made plastic pack measuring 2.5 X5 cm containing ice gel will be placed intraorally in the mouth on the vestibular surface of the treated tooth.
  Patients will be instructed to remove the ice pack for 2 minute if they felt extreme cold or a burning sensation. Each pack will be placed for 10 min, totaling three minimally per 30 min of intermittent application with 2-min breaks in between.
  During the cryotherapy treatment, a thermocouple device will be used to monitor the temperature, which Will be maintained at 10 °C. If the temperature exceeded the predetermined threshold of 10 °C, immediate replacement of the gel pack with a new one will be carried out to bring the temperature back within the desired range.
  Interventions: Procedure: oral Cryotherapy
- Intra-Radicular Cryo Group (Active Comparator): During the procedure, irrigation was performed between each rotary file using a side-vented needle (gauge size 30) positioned 2mm from the working length. This was done with 5 mL of 2.5% sodium hypochlorite (NaOCl), Followed by 5 ml of 17% EDTA (META BIOMED, Korea) for 1 min. Final flush was done with cold (2-4 oC) Saline for 10 mins.
  Interventions: Procedure: Intra radicular Cryotherapy
- Cold Irr. group (Active Comparator): Canals were irrigated with cold (2-4 oC) 2.5% NaOCl. Final flush was done with cold (2-4 oC) Saline for 10 mins.
  Interventions: Procedure: cold irrigation

INTERVENTIONS:
Procedure: oral Cryotherapy — custom made plastic pack measuring 2.5 X5 cm containing ice gel will be placed intraorally in the mouth on the vestibular surface of the treated tooth.
  Arms: Oral Cryo Group
Procedure: Intra radicular Cryotherapy — Final flush was done with cold (2-4 oC) Saline for 10 mins.
  Arms: Intra-Radicular Cryo Group
Procedure: cold irrigation — irrigation with cold (2-4 oC) 2.5% NaOCl and Final flush was done with cold (2-4 oC) Saline for 10 mins.
  Arms: Cold Irr. group

SUMMARY:
Pain is the major reason for patients' visits to dental clinics.Medications have side effects. Treatments including cryotherapy have been suggested to prevent these side effects.This study will compare the effect of oral and intraradicular cryotherapy on the level of substance p ,post operative pain and analgesic intake in mandibular premolars with symptomatic apical periodontitis.

Thirty patients with symptomatic apical periodontitis will be randomly distributed into three groups: oral,intraradicular cryotherapy and control group (n = 10). In the oral cryotherapy group application of (a cold pack of ice gel enveloped by a sealed plastic cover) will be performed for 30 minutes following the completion of canal preparation.Getting glide path by inserting K-file #10. coronal flaring will be done .The first apical fluid samples for all groups will be obtained at this step. Intra-radicular cryotherapy will be performed where normal root canal treatment will be done. Then a final flush will be done with 20 mL of cold saline 2.5°C for 10 minutes.

For the control group,no application of cryotherapy will be done.Second samples will be taken after mechanical preparation for intraradicular and control ,and after 30minutes of cold application for the cryotherapy group.Levels of substance p will be measured using the ELISA test.The patients will be asked to fill out the VAS questionnaire at 6, 24, 48 and 72 h.and analgesic intake

DETAILED DESCRIPTION:
-Oral Cryo Group: All patients will receive anesthesia containing Artinibsa 4%:100,000 epinephrine (Inibsa, Spain) 1.8 mL .

The teeth will be isolated with a rubber dam (Sanctuary) after local anesthesia. Dental caries or restoration of the teeth, if any, will be removed .Access cavity will be done by new tapered stone with round end with copious coolant. Upon pulp exposure, dark profuse bleeding filled the pulp chamber. Initial glide path will be done by inserting K-file #10. After confirming glide path, coronal flaring will be done by orifice opener rotary file (M-Pro 19 taper 8). Working length will be determined by apex locator E PEX (Eighteeth Medical Technology Co., Ltd., Changzhou, China).The working length will be established at 0.5 mm short of the full length as determined by the electronic apex locatorand validated by a periapical radiograph.

First base line apical fluid sample (S1) will be collected at this step. Sterile paper point size 20 taper 2% will be inserted into the canal and placed 2 mm beyond the apex. The paper point will be left for 30 seconds to absorb sufficient amount of fluid. Paper point will be placed into an Eppendorf tube with 1 mL (pH 7.4) phosphate buffered saline and refrigerated at 10°C for later examination.

Mechanical preparation of the canals will be carried out according to the sequence of M pro rotary files kit #20/4, #25/6, #35/4, #40/4. Patency will be checked after each file with #10 k- file. Apical preparation will be further enlarged to manual file #50 or #55 in some cases. During the procedure, irrigation will be performed between each rotary file using a side-vented needle (gauge size 30) positioned 2mm from the working length. This will be done with 5 mL of 2.5% sodium hypochlorite (NaOCl). Followed by 5 ml of 17% EDTA (META BIOMED, Korea) for 1 min.Final flush will be done with room temperature Saline for 10 minutes.

Next, custom made plastic pack measuring 2.5 X5 cm containing ice gel will be placed intraorally in the mouth on the vestibular surface of the treated tooth.

Patients will be instructed to remove the ice pack for 2 minute if they felt extreme cold or a burning sensation. Each pack will be placed for 10 min, totaling three minimally per 30 min of intermittent application with 2-min breaks in between.

During the cryotherapy treatment, a thermocouple device will be used to monitor the temperature, which Will be maintained at 10 °C. If the temperature exceeded the predetermined threshold of 10 °C, immediate replacement of the gel pack with a new one will be carried out to bring the temperature back within the desired range.

After the completion of three cycles, the second sample of AF (S2) will be collected, as described earlier.

-Intra-Radicular Cryo Group: Access cavity was done by new tapered stone with round end with copious coolant. Upon pulp exposure, dark profuse bleeding filled the pulp chamber. Caries and old restoration were removed.

Initial glide path was done by inserting K-file #10. After confirming glide path, coronal flaring was done by orifice opener rotary file (M-Pro 19 taper 8). Working length was determined by apex locator.

First base line apical fluid sample (S1) was collected at this step. Sterile paper point size 20 taper 2% was inserted into the canal and placed 2 mm beyond the apex. The paper point was left for 30 seconds to absorb sufficient amount of fluid.

Mechanical preparation of the canals was carried out according to the sequence of M pro rotary files kit #20/4, #25/6, #35/4, #40/4. Patency was checked after each file with #10 k- file. Apical preparation was further enlarged to manual file #50 or #55 in some cases.

During the procedure, irrigation was performed between each rotary file using a side-vented needle (gauge size 30) positioned 2mm from the working length. This was done with 5 mL of 2.5% sodium hypochlorite (NaOCl), Followed by 5 ml of 17% EDTA (META BIOMED, Korea) for 1 min. Final flush was done with cold (2-4 oC) Saline for 10 mins. Temperature of cold saline was maintained by keeping the irrigation syringes in an ice box filled with cooling gel packs with thermocouple inside to confirm that the temperature within range (2-4 oC). Irrigation syringes were used one by one.

The second sample (S2) was taken after chemo-mechanical preparation and finishing the irrigation protocol.

Cold Irrigation Group :

Canals were irrigated with cold (2-4 oC) 2.5% NaOCl. Final flush was done with cold (2-4 oC) Saline for 10 mins. First apical fluid sample will be taken after coronal flaring and determining the working length and the second one was taken after chemo-mechanical preparation and finishing the irrigation protocol.

-Control Group: Patients will receive conventional root canal treatment. Canals will be irrigated with room temperature 2.5% NaOCl. Final flush will be done with room temperature saline for 10 min.First apical fluid sample will be taken after coronal flaring and determining the working length and the second one was taken after chemo-mechanical preparation and finishing the irrigation protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Eligible participants will be between the ages of 18-45
3. Participants willing to commit for the entire period of the trial and agreed to sign the written consent after full explanation of the study
4. Having a mandibular single rooted premolar tooth with vital pulp Vertucci Type I canal system.
5. Patients that will be diagnosed with symptomatic apical periodontitis on the basis of the clinical symptoms of severe preoperative pain (visual analogue scale [VAS] > 7) and severe percussion pain (VAS > 7)
6. The absence of periapical radiolucency on x ray.

Exclusion criteria :

1. Presence of any systemic disease or allergic reactions
2. Vulnerable population: prisoners, pregnant women, mentally ill people, etc.
3. Use of analgesic or antibiotic medication within seven days
4. A radiographically untraceable canal
5. Excessively curved root
6. Excessively long or short root length
7. Teeth with open apices
8. A previous root canal treatment
9. Sinus tracts
10. Local gum swelling around the affected tooth
11. Severe periodontal disease
12. Presence of periodontal pockets >3 mm in the affected tooth
13. Absence of bleeding in the pulp chamber on access cavity preparation
14. Problems in determining working length
15. Broken files, over instrumentation, and overfilling/incomplete filling

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Level of inflammatory mediator (substance P) in apical fluid | base line 1st sample:after glide path and coronal flaring for all groups second sample:in control group and intraradicular group taken after mechanical preparation, ,and in oral cryo group after mechanical application and 30 minutes application of cryo
  Sterile paper point size 20 taper 2% will be inserted into the canal and placed 2 mm beyond the apex. The paper point will be left for 30 seconds to absorb sufficient amount of fluid. Paper point will be placed into an Eppendorf tube with 1 mL (pH 7.4) phosphate buffered saline and refrigerated at 10°C for later examination.After collecting samples from all patients, the samples will be evaluated by the enzyme-linked immunosorbent assay (ELISA) method.

SECONDARY OUTCOMES:
level of post operative pain using 10 cm visual analoge scale (VAS) | after 6hours, 24hours, 48hours, 72hours h after treatment
  On a10-cm Visual Analogue Scale (VAS) questionnaire, each patient reported their level of pain as follows: There is no pain at 0, 1-3, mild, 4-6, moderate, 7-9, severe, and 10, the worst pain
Analgesic intake | They will be contacted by telephone at 6, 12, 24, 48 and 72 hours after
  They will be asked if they needed to take the analgesics and the frequency of taking it.

CONTACTS AND LOCATIONS:
Overall Officials: Maram F Obeid, Professor, Study Director — Faculty of Dentistry,Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Detailed study protocol
Supporting Information: Study Protocol
Time Frame: 2027,for a year
Access Criteria: review purpose of request,

REFERENCES:
- [Background] Abdel-Baset ST, Fahmy SH, Obeid MF. Can instrumentation kinematics affect postoperative pain and substance P levels? A randomized controlled trial. BMC Oral Health. 2024 Jan 17;24(1):102. doi: 10.1186/s12903-024-03882-x. PMID 38233887
- [Background] Sharaf RMA, Abdelrahman TY, Obeid MF. The impact of using cold irrigation on postoperative endodontic pain and substance P level: a randomized clinical trial. Odontology. 2025 Jun 18. doi: 10.1007/s10266-025-01131-3. Online ahead of print. PMID 40533695
- [Background] Hamza EM, Abd El Aziz TM, Obeid MF. The influence of intraoral cryotherapy on postoperative pain and substance P in symptomatic apical periodontitis: randomized clinical study. Sci Rep. 2024 Jun 17;14(1):13890. doi: 10.1038/s41598-024-64071-y. PMID 38880787
- [Background] Vera J, Ochoa J, Romero M, Vazquez-Carcano M, Ramos-Gregorio CO, Aguilar RR, Cruz A, Sleiman P, Arias A. Intracanal Cryotherapy Reduces Postoperative Pain in Teeth with Symptomatic Apical Periodontitis: A Randomized Multicenter Clinical Trial. J Endod. 2018 Jan;44(1):4-8. doi: 10.1016/j.joen.2017.08.038. Epub 2017 Nov 1. PMID 29079057